CLINICAL TRIAL: NCT03432494
Title: Early Feasibility Evaluation of Transmural Systems Transcaval Closure Device (TCD) for Transcaval Access Ports During Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: Transmural Systems Transcaval Closure Device for Transcaval Access Ports During Transcatheter Aortic Valve Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was kept open (via administrative hold) in anticipation of a device redesign and enrollment suspended, but funding never materialized to support the redesign.
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 999918045; 18-H-N045
Record Dates: First submitted 2018-02-13; First posted 2018-02-14 (Actual); Results first posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-03

CONDITIONS: Aortic Stenosis
Keywords: Transcatheter; Transcaval; Bioprosthesis; Closure Device; Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Transcaval access and closure with the transcaval closure device (TCD) test article. (Experimental): All participants undergo transcaval access for transcatheter aortic valve replacement (TAVR) followed by implantation of the transcaval closure device (TCD).
  Interventions: Device: Transcaval closure device (TCD)

INTERVENTIONS:
Device: Transcaval closure device (TCD) — Transcaval access and closure using the Transmural Transcaval Closure Device (TCD) at the time of medically-necessary transcatheter aortic valve replacement (TAVR).

SUMMARY:
Background:

Transcatheter aortic valve replacement (TAVR) is a non-surgical alternative to standard surgical aortic valve replacement. Not all patients are eligible for TAVR using standard access through the artery in the groin, because the artery is too small or too diseased. In this study, TAVR is performed using a new technique called transcaval access. The catheter is placed in the artery deep in the body by crossing through the wall of a deep vein. The connection between that vein and the aorta is closed with a new metallic device they are testing. This is called a transcaval closure device (TCD).

Objective:

To test the safety and early feasibility of closure of transcaval aortic access sites using the TCD after TAVR.

Eligibility:

Adults ages 21 and older undergoing TAVR for whom the procedure cannot be performed safely by the standard artery approach

Design:

Participants will be assessed by heart experts including cardiologists and surgeons.

Participants will have TAVR by the transcaval approach. A small catheter will be passed between the largest vein in the body and the nearby largest artery (aorta), inside the abdomen. Through this catheter, the TAVR will be implanted in the usual way.

After, doctors will implant the TCD by catheter to close the hole made in the aorta.

Participants will be X-rayed. A dye will be injected to view the TCD device.

Participants will get standard TAVR care afterwards. They will have physical exams, blood tests, and scans.

Participants will have a follow-up scan within 1 month and after 12 months.

Participants will have follow-up visits and phone calls 6 and 12 months after the procedure.

DETAILED DESCRIPTION:
Transcaval access to the abdominal aorta from the neighboring inferior vena cava (IVC) enables transcatheter aortic valve replacement (TAVR) in patients not eligible for femoral artery access. Currently the procedure is performed using devices, off-label, designed and marketed to close holes inside the heart and great vessels, manufactured by Abbott St Jude (Amplatzer Duct Occluder and Amplatzer Muscular VSD Occluder). Because these Amplatzer occluders are not designed to close transcaval access sites, they may not completely prevent bleeding.

This is an early feasibility study (EFS) evaluation of a purpose-built closure device for transcaval access. The device, the Transcaval closure device (TCD) will be evaluated for safety and performance to close transcaval access sites in patients ineligible for femoral artery access for TAVR.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Consents to participate in this study and all related clinical follow-up procedures
* Adults age greater than or equal to 21 years
* Undergoing transcatheter aortic valve replacement (TAVR) based on the clinical assessment of the multidisciplinary heart team
* Ineligible for femoral artery access for the selected transcatheter heart valve (THV) according to the THV manufacturer instructions for use. (Note Corevalve Evolut R: greater than or equal to 5mm; Evolut PRO 23, 26, 29 mm valves and Evolut R 34 mm: greater than or equal to 5.5 mm; Edwards Sapien 3, 23-26mm: 5.5 mm; Edwards Sapien 3, 29mm: 6.0mm; Anatomic ineligibility also considers patient-specific pattern of iliofemoral calcium and tortuosity.)
* Eligible for transcaval access based on Core lab analysis of the baseline abdomen/pelvis CT indicating a calcium-free target window on the abdominal aorta; a target greater than or equal to 15mm from the lowest main renal artery or aorto-iliac bifurcation; no important interposed structures; a projected intravascular centerline distance from the lower femoral head to the target at least 5cm less than the intended THV introducer sheath; patient celiac or superior mesenteric artery
* Aorta diameter greater than or equal to 11mm at the target crossing site
* Concordance of the study eligibility committee

EXCLUSION CRITERIA:

* High risk features on baseline CT including porcelain aorta (confluent calcification); pedunculated aortic atheroma; or leftward aortic angel greater than or equal to 20 degrees with regard to vertical.
* Renal dysfunction limiting follow-up contrast-enhanced CR (estimated glomerular filtration rate, eGFR less than 30mL/min/1.73m^2 if not already on renal replacement therapy)
* Pregnancy or intent to become pregnant prior to completion of all protocol follow-up procedures

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Lederman, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (3):
- United States (3):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Henry Ford Hospital, Detroit, Michigan

IPD SHARING:
Plan to Share IPD: No
The authors are willing to share de-identified subject data upon reasonable request

REFERENCES:
- [Derived] Rogers T, Greenbaum AB, Babaliaros VC, Stine AM, Khan JM, Schenke WH, Eng MH, Paone G, Leshnower BG, Satler LF, Waksman R, Chen MY, Lederman RJ. Dedicated Closure Device for Transcaval Access Closure: From Concept to First-in-Human Testing. JACC Cardiovasc Interv. 2019 Nov 11;12(21):2198-2206. doi: 10.1016/j.jcin.2019.05.053. Epub 2019 Oct 16. PMID 31629746

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Started | 12
Completed | 10
Not Completed | 2
Not completed — Death | 1
Not completed — Noncompliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 12
Ineligible for transfemoral access [Count of Participants; unit: Participants] | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Technical Success of Delivery of the Transcaval Closure Device (TCD)
Description: Number of participants with technical success of delivery of the transcaval closure device (TCD)
  All of the following must be present for technical success:
  1. Alive
  2. Successful delivery of the TCD, and retrieval of the TCD delivery system
  3. Deployment and correct positioning of a single intended TCD. Repositioning and recapture of the device, if needed, is not classified as failure.
  4. No additional unplanned or emergency surgery or re-intervention related to the TCD or delivery system
  5. Adjunctive balloon aortic tamponade is permissible and consistent with technical success
Time Frame: 1 minute following procedure discharge (Exit from the catheterization laboratory)
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 12

2. Secondary Outcome: Number of Participants With Closure Success of the Transcaval Closure Device (TCD)
Description: Number of Participants With Technical Closure Success of Delivery of the Transcaval Closure Device (TCD). This secondary endpoint is a composite of the primary endpoint and hemostasis of the transcaval aortic access site.
  All of the following must be present for Closure Success:
  1. Alive
  2. Successful delivery of the TCD, and retrieval of the TCD delivery system
  3. Deployment and correct positioning of a single intended TCD. Repositioning and recapture of the device, if needed, is not classified as failure.
  4. No additional unplanned or emergency surgery or re-intervention related to the TCD or delivery system. Adjunctive balloon aortic tamponade is permissible and consistent with technical success
  5. Complete occlusion of the aortocaval fistula on the completion aortogram.
Time Frame: 1 minute following procedure discharge (Exit from the catheterization laboratory)
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 9

3. Secondary Outcome: Number of Participants Who Experienced Device Success of the Transcaval Closure Device (TCD)
Description: A key performance endpoint is the number of participants who experienced device success of the transcaval closure device (TCD).
  All of the following must be present for device success:
  1. Alive or Death unrelated to transcaval access or TAVR
  2. Original intended TCD in place
  3. No additional surgical or interventional procedures related to access or the device after exit from the cath lab
  Intended performance of the TCD, including all of:
  1. Structural Performance: No migration, embolization, detachment, fracture, hemolysis, or endarteritis related to the TCD
  2. Hemodynamic performance: No abdominal aortic obstruction caused by the TCD implant
  3. Absence of para-device complications (large retroperitoneal hematoma, pseudoaneurysm, distal thromboembolism, or pulmonary thromboembolism)
Time Frame: 30 days and 12 Months
Population: Data will be analyzed using principles both of (1) intention-to-treat, defined as attempting or initiating transcaval crossing procedures, and (2) as-treated, defined as completing transcaval closure attempts.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  30 Days | 12
  12 Months: number analyzed (Participants) | 10
  12 Months | 10

4. Secondary Outcome: Number of Participants That Experienced Procedural Success
Description: Number of participants that experienced safety endpoint of procedural success following transcaval closure device (TCD) at day 30.
  All of the following must be present for procedural success:
  1. Device success
  2. No device-related Serious Adverse Events, defined as VARC-2 life-threatening bleeding, major vascular or cardiac complications related to the TCD requiring unplanned reintervention or surgery (such as covered stent implantation at the transcaval access site)
Time Frame: 30 Days
Population: Intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 12

5. Secondary Outcome: Number of Participants Requiring Covered Stent Implantation as a Normal Provisional Part of the Procedure
Description: Number of participants requiring covered stent implantation as a normal provisional part of the procedure assessed during the procedure.
Time Frame: During procedure, procedure may last from 2 to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 0

6. Secondary Outcome: Number of Participants With Covered Stent Implantation at the Transcaval Closure Device Implantation Site
Description: Number of participants with covered stent implantation at the transcaval closure device (TCD) implantation site
Time Frame: During procedure, procedure may last from 2 to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 0

7. Secondary Outcome: Number of Participants Final Acute Aorto-caval Fistula Score
Description: Number of Participants final acute aorto-caval fistula score at procedure completion.
  Scoring is defined as: Type 0=occlusion, Type 1=patent fistula, Type 2=cruci-form fistula pattern, Type 3=extravasation.
  A score of 0 is associated with complete occlusion at the transcaval closure device (TCD) site while a higher score is associated with incomplete occlusion at the TCD site.
Time Frame: 30 Days
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Type 0 | 9
  Type 1 | 1
  Type 2 | 2
  Type 3 | 0

8. Secondary Outcome: Number of Participants Who Experienced Modified Valve Academic Research Consortium-2 Vascular Complications
Description: Participants who experienced Minor or Major modified Valve Academic Research Consortium-2 (VARC-2) vascular complications.
  Major is defined as: Aortic dissection or aortic rupture; Access site-related arterial or venous injury THAT RESULTS IN death, hemodynamic compromise, life-threatening, extensive; or major bleeding, visceral ischemia, neurological impairment; Distal embolization requiring surgery or resulting in amputation or irreversible end-organ damage; severe access site vascular complication Minor is defined as: Access site-related arterial or venous injury THAT DOES NOT RESULT IN death, hemodynamic compromise, life-threatening, extensive; or major bleeding, visceral ischemia, neurological impairment; Distal embolization treated with embolectomy and/or thrombectomy not resulting in amputation or irreversible end-organ damage; Any unplanned endovascular stenting or unplanned surgical intervention not meeting the criteria for a major vascular complication; Vascular repair
Time Frame: 30 days
Population: intention-to-treat (ITT) analysis
Measure: Number; unit: participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
participants
  Major : Unrelated to Transcaval Closure Device | 0
  Major : At Least Possibly Related to Transcaval Closure Device | 0
  Minor Unrelated to Transcaval Closure Device : Unrelated to Transcaval Closure Device | 1
  Minor Unrelated to Transcaval Closure Device: At Least Possibly Related to Transcaval Closure Device | 1

9. Secondary Outcome: Number of Participants Who Experienced Modified Valve Academic Research Consortium-2 Bleeding Complications
Description: Number of Participants Who Experienced Major or Life-threatening Modified Valve Academic Research Consortium-2 (VARC-2) bleeding complications at 30 days
  Major defined as: Corrected drop in the hemoglobin of >=3.0 g/dl AND does not meet criteria of life-threatening or extensive bleeding; Requiring transfusion of >=3 U of whole blood or packed RBCs AND does not meet criteria of life-threatening or extensive bleeding.
  Life-threatening defined as: Intracranial requiring surgery or intervention; Intraspinal requiring surgery or intervention; Intraocular requiring surgery or intervention; Pericardial requiring surgery or intervention; Intramuscular with compartment syndrome; Bleeding causing hypovolemic shock or hypotension or requiring significant doses of vasopressors or surgery
Time Frame: 30 Days
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Life-threatening : Unrelated to Transcaval Closure Device | 0
  Life-threatening : At least Possibly Related to Transcaval Closure Device | 0
  Major : Unrelated to Transcaval Closure Device | 1
  Major : At least Possibly Related to Transcaval Closure Device | 0

10. Secondary Outcome: Number of Participants Who Experienced Major Adverse Cardiovascular Events
Description: Number of Participants Who Experienced Major Adverse Cardiovascular Events (MACE)
  Major adverse cardiovascular events (MACE), defined as VARC-2 Early Safety composite: No mortality, stroke, life-threatening bleeding, acute kidney injury (AKI) stage 2+, major vascular complication, and valve-related complication.
Time Frame: Day 30
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Stroke : Unrelated to Transcaval Closure Device | 2
  Stroke : At least possibly related to Transcaval Closure Device | 0
  Myocardial Infraction : Unrelated to Transcaval Closure Device | 1
  Myocardial Infraction : At least possibly related to Transcaval Closure Device | 0
  Acute Kidney Injury (Stage II or III) : Unrelated to Transcaval Closure Device | 0
  Acute Kidney Injury (Stage II or III) : At least possibly related to Transcaval Closure Device | 0

11. Secondary Outcome: Number of Participants With Closure Success of Delivery of the Transcaval Closure Device (TCD)
Description: Number of Participants With Closure Success of Delivery of the Transcaval Closure Device (TCD).
  All of the following must be present for Closure Success:
  1. Alive or Death unrelated to transcaval access or TAVR
  2. Successful delivery of the TCD, and retrieval of the TCD delivery system
  3. Deployment and correct positioning of a single intended TCD. Repositioning and recapture of the device, if needed, is not classified as failure.
  4. No additional unplanned or emergency surgery or re-intervention related to the TCD or delivery system. Adjunctive balloon aortic tamponade is permissible and consistent with technical success
  5. Complete occlusion of the aortocaval fistula on the completion aortogram.
Time Frame: 30 Days and 12 Months
Population: Data will be analyzed using principles both of (1) intention-to-treat, defined as attempting or initiating transcaval crossing procedures, and (2) as-treated, defined as completing transcaval closure attempts. For 12 months analysis, one participant died and one participant taken off study due to noncompliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  30 Days | 12
  12 Months: number analyzed (Participants) | 10
  12 Months | 10

12. Secondary Outcome: All-Cause Mortality
Description: All-cause mortality, as categorized by cardiovascular vs non-cardiovascular, peri- vs non-periprocedural, regardless of attribution to Transcaval Closure Device (TCD)
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Cardiovascular Deaths : Unrelated to Transcaval Closure Device | 0
  Cardiovascular Deaths : At least possibly related to Transcaval Closure Device | 0
  Non-Cardiovascular Deaths : Unrelated to Transcaval Closure Device | 1
  Non-Cardiovascular Deaths : At least possibly related to Transcaval Closure Device | 0

13. Secondary Outcome: Number of Participants With Aorto-caval Fistula Patency Assessed by Angiography and Arterial-phase Follow-up Computed Tomography
Description: Number of participants with aorto-caval fistula patency at each timepoint, assessed combining completion angiography and arterial-phase follow-up Computed tomography (CT).
Time Frame: Day 30, 12 months
Population: Data will be analyzed using principles both of (1) intention-to-treat, defined as attempting or initiating transcaval crossing procedures, and (2) as-treated, defined as completing transcaval closure attempts. For month 12, one participant died and one participant taken off study due to noncompliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Day 30 | 12
  12 Months: number analyzed (Participants) | 10
  12 Months | 10

14. Secondary Outcome: Number of Participants Who Experienced Acute Kidney Injury Stage 2 or 3
Description: Number of participants who experienced acute kidney injury (AKI) stage 2 or 3 using the Valve Academic Research Consortium (VARC).
  AKI using the VARC definition:
  Stage 2: increase in serum creatinine to 200-300% (2.0-3.0 times increase compared to baseline) or increase of >0.3 mg/dl (>26.4 mmol/L) but <4.0 mg/dl (<354 mmol/L)
  Stage 3: increase in serum creatinine to ≥300% (>3 times increase compared to baseline) or serum creatinine of ≥4.0 mg/dl (≥354 mmol/L), with acute increase of ≥0.5 mg/dl (44 mmol/L)
Time Frame: 30 Days
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Acute Kidney Injury, Stage II | 0
  Acute Kidney Injury, Stage III | 0

15. Secondary Outcome: Number of Participants That Are Free From Infection Related to the Transcaval Closure Device
Description: Number of participants that experience freedom from infection related to the Transcaval Closure Device (TCD) at each time point
Time Frame: Day 30, 12 Months
Population: Intention-to-treat (ITT) analysis. One participant died on post-procedure day 15 from respiratory failure attributed to exacerbation of previously unrecognized fibrotic pulmonary disease, adjudicated as noncardiovascular mortality and unrelated to transcaval access or TAVR. One participant at month 12 was taken off study due to non-compliance.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Day 30 | 12
  12 months: number analyzed (Participants) | 10
  12 months | 10

16. Secondary Outcome: Number of Participants That Experience Thrombocytopenia and is Attributable to Residual Aorto-caval Fistula or the Transcaval Closure Device
Description: Number of participants that experience Thrombocytopenia as defined as < 50,000 and is attributable to residual aorto-caval fistula or the Transcaval Closure Device (TCD)
Time Frame: 30 Days
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 0

17. Secondary Outcome: Number of Participants Who Experience Hemolysis and is Attributable to Residual Aorto-caval Fistula or the Transcaval Closure Device
Description: Number of participants who experience hemolysis and is attributable to residual aorto-caval fistula or the Transcaval Closure Device (TCD)
Time Frame: 30 Days
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 1

18. Secondary Outcome: Participant Cumulative Computed Tomography Analysis of Device
Description: Participant cumulative Computed tomography (CT) analysis of device. As defined by: Device position; Device integrity; Aortocaval tract pseudo-aneurysm; Aortic pseudoaneurysm; Retroperitoneal hematoma grade (stranding {=absent and not evidence of overt bleeding;} small; moderate; larger); Intracaval mass or thrombus; Aortic dissection and inferred relatedness to TCD (adjacent to access port) or procedure (remote to access port)
Time Frame: Day 30
Population: intention-to-treat (ITT) analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants
  Migration | 0
  Erosion | 0
  Retroperitoneal hematoma | 0
  Aortic pseudoaneurysm | 0
  Aortocaval tract pseudo-aneurysm | 0
  Intracaval mass or thrombus | 0
  Aortic dissection | 0

19. Secondary Outcome: Number of Participants Enrolled Greater Than 65 Years
Description: Outcomes of subjects greater than 65 years (i.e. eligible for Medicare based on age), to determine generalizability to the Medicare population
Time Frame: Enrollment
Population: One participant is under 65 years of age and not included.
Measure: Count of Participants; unit: Participants
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
Number analyzed (Participants) | 12
Participants | 11

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events and adverse device effects will captured up to day 30 follow up, then only serious adverse events (SAE), serious adverse device effects (SADE), unanticipated de-vice effects (UADE) and unanticipated problems (UP) will be reported for remainder of study (12 month follow up).
Arm/Group | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article
All-Cause Mortality (participants affected / at risk) | 1/12
Serious Adverse Events (participants affected / at risk) | 9/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac Chest pain (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Mobitz (type) II atrioventricular block (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
C. Difficile infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Stroke (Nervous system disorders) | 2 (3)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Arterial thromboembolism (Vascular disorders) | 1 (1)
Labile blood pressure (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transcaval Access and Closure With the Transcaval Closure Device (TCD) Test Article (N=12)
Anemia (Blood and lymphatic system disorders) | 12 (12)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 7 (7)
Aortic valve disease (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Mild AVR paravalvular leak (Cardiac disorders) | 1 (1)
Moderate PV aortic regurgitation (Cardiac disorders) | 1 (1)
Cardiac Chest pain (Cardiac disorders) | 2 (2)
Conduction disorder (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (2)
Left femoral hematoma (Injury, poisoning and procedural complications) | 1 (1)
Right groin oozing (Injury, poisoning and procedural complications) | 1 (1)
Small right groin hematoma (Injury, poisoning and procedural complications) | 1 (1)
Head laceration with fall (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 9 (9)
Cardiac troponin I increased (Investigations) | 10 (10)
Creatinine increased (Investigations) | 3 (5)
Haptoglobin decreased (Investigations) | 2 (2)
Elevated BNP (Investigations) | 3 (3)
Elevated BUN (Investigations) | 1 (1)
Elevated Haptoglobin (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 6 (6)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
In-situ squamous cell carcinoma lesion on right dorsal forearm. (Skin and subcutaneous tissue disorders) | 1 (1)
Arterial thromboembolism (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The clinical trial was put suspended due to device needing to be redesign however funding never materialized to support the redesign, therefore, clinical trials was terminated early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT03432494/Prot_SAP_000.pdf